CLINICAL TRIAL: NCT05989893
Title: Mapping of Human Cognition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Nitin Tandon, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-06-0385; U01NS128921 (NIH)
Record Dates: First submitted 2023-07-27; First posted 2023-08-14 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy; Brain Tumor
Keywords: seizure
MeSH Terms: conditions — Epilepsy; Brain Neoplasms; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neural recordings and stimulation during language tasks (Experimental)
  Interventions: Behavioral: Language-based tasks

INTERVENTIONS:
Behavioral: Language-based tasks — In either the MRI suite, or the Epilepsy Monitoring Unit, or the operating room, epilepsy and tumor subjects are asked to perform a variety of language-based tasks as neural recordings are made from and/or neural stimulations are delivered to various language areas of the brain.

SUMMARY:
The purpose of this study is to compare organization of normal brain function as detected using Functional magnetic resonance imaging (fMRI) in normal subjects as opposed to patients with epilepsy or brain tumors, to ascribe precise anatomic labels (including Brodmann Areas) and functional significance to each region involved in cognitive processes as detected by cortical stimulation mapping (CSM) in patients with implanted subdural electrodes (SDE) or depth (sEEG) electrodes, to describe the locations of these regions in Talairach space, for a population of patients without overt structural abnormalities in these regions, to generate a spatial probability map of locations of cortical regions "essential" for these processes, to compare the loci of "crucial" language, visual, motor and cognitive sites as determined by CSM with the loci determined by a battery of tasks using fMRI for each individual and to use these data in patients undergoing intracranial electro-corticographyto determine the loci of essential, involved and uninvolved brain areas, and use sophisticated mathematical analyses of these intracranial recordings to study information flow between these areas.

ELIGIBILITY:
Inclusion Criteria:

* patients with medically refractory epilepsy who are scheduled to undergo or have previously undergone placement of sub-dural electrodes (including depth electrodes) to localize the site of seizure onset and to map the locations of critical language and motor regions
* patients with epilepsy, brain tumors or cortically based vascular malformations (cavernous malformations or arterio-venous malformations) with lesions that are/were proximate to crucial brain regions, and who are scheduled to undergo or have previously undergone intra-op mapping of motor, visual or language function, or a Wada test, or maybe part of an awake craniotomy.
* proficiency in English

Exclusion Criteria:

* Gross structural abnormalities (large hamartomata, tumors, large vascular malformations, very large diffuse malformations of cortical development) that may have impacted upon the location of critical brain areas.
* Unable to participate in testing due to impaired cognition or mental retardation.
* Cardiac pacemakers, intracranial aneurysm clips, or other potentially mobile implanted metallic devices
* Patients with claustrophobia who cannot undergo an MRI scan without sedation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in reading errors as assessed by the number of words read incorrectly | Baseline, during stimulation( about 2 seconds after baseline )
Change in reaction times in milliseconds | Baseline, during stimulation( about 2 seconds after baseline )
  reaction time is the time it takes to say the word after seeing it

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Tandon, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No